CLINICAL TRIAL: NCT01891890
Title: Cognitive AED Outcomes in Pediatric Localization Related Epilepsy (COPE)
Acronym: COPE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Emory University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, David Loring, PhD, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00066541; PCORI 527 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Results first posted 2017-09-19 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-07

CONDITIONS: Epilepsy, Partial; Epilepsy, Localization Related
Keywords: Pediatrics
MeSH Terms: conditions — Epilepsies, Partial | interventions — Oxcarbazepine; Levetiracetam; Lamotrigine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lamotrigine (Active Comparator): Lamotrigine 7.0 mg/kg tablets or chewable tablets administered daily in 2 equally divided doses
  Interventions: Drug: Lamotrigine
- Oxcarbazepine (Active Comparator): Oxcarbazepine 25 mg/kg tablets or liquid administered daily in 2 equally divided doses
  Interventions: Drug: Oxcarbazepine
- Levetiracetam (Active Comparator): Levetiracetam 30 mg/kg tablet or liquid administered daily in 2 equally divided doses
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Oxcarbazepine — Titration to target dose starting at week 3. Dose increments above target may be made to a maximum of 3 increments with a minimum interval between dose escalations of 2 weeks.
  Other Names: Trileptal
  Arms: Oxcarbazepine
Drug: Levetiracetam — Titration to target dose starting at week 3. Dose increments above target may be made to a maximum of 3 increments with a minimum interval between dose escalations of 2 weeks.
  Other Names: Keppra
  Arms: Levetiracetam
Drug: Lamotrigine — Titration to target dose starting at week 11. Dose increments above target may be made to a maximum of 3 increments with a minimum interval between dose escalations of 2 weeks.
  Other Names: Lamictal
  Arms: Lamotrigine

SUMMARY:
Seizures that arise in specific areas in the brain are called Localization Related Epilepsy (LRE) and are the most common seizure disorder in children. Children that receive drug treatment for this disorder may suffer from treatment related side effects which impact their ability to think or concentrate and their ability to interact socially. These negative treatment effects can impact the child's performance in school and long term may impact employment and job options.

This study will determine whether changes in attention and social interactions are seen in children treated for LRE using three of the most common medications used to treat pediatric LRE. Children who are newly diagnosed with LRE by their doctors and are between the ages of 5 years 6 months and 16 years 0 months will be randomized to receive levetiracetam, lamotrigine, or oxcarbazepine.

There will be 14 study sites throughout the US. Children will undergo evaluation of their thinking and ability to pay attention before and after starting drug treatment for LRE. Regardless of the specific findings, results of this study will provide the information needed to help parents and their clinicians choose treatment options that maximize cognitive abilities in children with LRE, and provide the data needed for practice guidelines to be established on the basis of cognitive side effect risks.

DETAILED DESCRIPTION:
This is a prospective multicenter, randomized, open-label, central assessor, parallel-group study of children ages 5 years, 6 months to 16 years, 0 months with newly diagnosed Localization Related Epilepsy (LRE) to establish whether three common antiepileptic drugs (AEDs) used as first line LRE treatment (lamotrigine (LTG), levetiracetam (LEV), or oxcarbazepine (OXC)) are associated with differential cognitive side effects on attention. It is predicted that one AED will be identified with greater negative cognitive effects on attention. The study will also examine whether there are differential risks for drug-related behavior change. The study will address whether 6 month attentional outcomes can be reliably predicted based upon shorter term cognitive change assessed soon after beginning AED therapy, and establish practice effects associated with repeated test exposure when on constant doses of AED.

Children will undergo cognitive testing after study enrollment and no more than a week after AED initiation. Selected measures will be repeated at the first follow up clinic visit after beginning AED treatment, and the primary endpoint will be the attention performance obtained at the subjects' 6 month follow-up clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Age of participant between 5 years, 6 months and 16 years, 0 months at the time of enrollment
* Weight is between ≥ 15 kg the lower limit BMI 99th percentile at study entry at study entry
* Child has diagnosed epilepsy as defined by one of the following definitions :

  * At least two unprovoked seizures occurring more than 24-hours apart, or
  * One unprovoked seizure and a probability of further seizures similar to the general recurrence risk after two unprovoked seizures (approximately 75% or more), or
  * At least two seizures in a setting of reflex epilepsy
* Child has a diagnosis of Localization Related Epilepsy (LRE) with or without secondary generalization according to International League Against Epilepsy (ILAE) criteria and which may include Benign Rolandic Epilepsy and Benign Occipital Epilepsy or other LREs.
* Localization related seizures will be based upon at least one of the following: 1) focal EEG abnormalities (sharp waves, spikes, or slowing) and the absence of generalized spike waves discharges, 2) focal MRI abnormalities other than active cysticercosis, which may include temporal lobe sclerosis, dysembryoplastic neuroepithelial tumor , ganglioglioma, or focal malformations of cortical development, 3) focal neurologic abnormalities, or 4) clinical semiology, which may include Todd's phenomenon, unilateral dystonia, or fencing posture, or distinct aura consistent with localization related seizure onset (e.g., classic déjà vu or bad smell).
* Participants must either be antiepileptic drug (AED) therapy naïve or on an AED (excluding benzodiazepines) for 1-week or less. Children may be on a stable dose of psychostimulants at the time of enrollment, but no change in medication, dose, or schedule in 3 months prior to study enrollment, with no anticipated dosing changes during the 6 months of the study. If participants are taking psychostimulants at the time of study entry, they should plan on continuing them for the 6 month duration of the study protocol including the 3-month and 6-month cognitive and behavioral testing time points.
* Females of child bearing potential must agree to acceptable forms of birth control, which may include abstinence.
* The child's parent/guardian must be able to keep an accurate seizure diary and be able and willing to comply with instructions and study procedures.
* Informed consent from the child's legal guardian or legal representative.
* Assent will be obtained from children according to each site's institutional guidelines.

Exclusion Criteria:

* Children with history of primary generalized seizures (absence, myoclonic, drop)
* Children with mixed seizure disorder (e.g., Lennox-Gastaut Syndrome)
* Children with sensory seizures only (i.e., auras)
* Children with 6+ seizures in the previous week
* Children with a history of status epilepticus
* Children with a history of neonatal seizures
* Children with diagnoses of pervasive developmental disorders (e.g., autism/autism spectrum disorders)
* Children with progressive neurological disease (e.g., degenerative, progressive neoplasm)
* Children with major medical disease (e.g., Insulin-Dependent Diabetes Mellitus (IDDM), cancer, renal failure)
* Children with diseases with cognitive impact (e.g., inborn errors of metabolism, sickle cell disease with history of stroke)
* Children with active cysticercosis documented on MRI
* Children with cognitive impairment of sufficient severity that, in the opinion of the investigator, would diminish the likelihood of valid test performance (roughly corresponding to Full Scale Intelligence Quotient (FSIQ) less than 70)
* Children with suicide attempt(s) at any point during their lifetime
* Children with active suicide ideation
* Children with chronic use of first generation antihistamines
* Children using recreational drugs (including alcohol)
* Children not fluent in either English or Spanish
* Female children who are pregnant
* Female children who are using oral contraceptives for birth control or for any other indication (e.g. acne treatment)

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2013-08; Primary Completion 2015-10-23 (Actual); Study Completion 2015-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W. Loring, PhD, Principal Investigator — Emory University
Locations (14):
- United States (14):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of California at San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healtcare of Atlanta, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - University of Rochester, Monroe, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 14 pediatric practices in the United States of America between August 2013 and October 2015.
Pre-assignment Details: In total, 78 individuals consented to participate in the trial. Of these 6 were found to be ineligible or declined to participate prior to receiving the intervention, resulting in 72 participants who received the study intervention.
Groups:
- Lamotrigine: Participants who received lamotrigine 7.0 mg/kg tablets or chewable tablets daily, administered in 2 equally divided doses
- Oxcarbazepine: Participants who received oxcarbazepine 25 mg/kg tablets or liquid daily, administered in 2 equally divided doses
- Levetiracetam: Participants who received levetiracetam 30 mg/kg tablet or liquid daily, administered in 2 equally divided doses
Period: Overall Study
Arm/Group | Lamotrigine | Oxcarbazepine | Levetiracetam
Started | 24 | 27 | 21
Completed | 17 | 24 | 14
Not Completed | 7 | 3 | 7
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Study ended before endpoint reached | 7 | 3 | 6

BASELINE CHARACTERISTICS:
Population: Patients who were eligible to participate and were randomized to a study arm are included in the baseline description.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lamotrigine | Oxcarbazepine | Levetiracetam | Total
Number analyzed (Participants) | 24 | 27 | 21 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 27 | 21 | 72
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.6 (2.0) | 8.6 (2.4) | 9.1 (2.1) | 8.7 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 11 | 36
  Male | 11 | 15 | 10 | 36
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 27 | 21 | 72

OUTCOME MEASURES:

1. Primary Outcome: Conners' Continuous Performance Test II (CPT-II) Confidence Index
Description: The Conners' Continuous Performance Test II (CPT-II) is a measure of sustained attention. Letters are individually presented on a computer screen, and participants are instructed to press the space bar when they are presented with any letter except the letter "X". For children younger than 6 years of age at enrollment, the Kiddie CPT will be used in which the child is instructed to press the space bar every time the ball appears on the screen. The outcome measure is a confidence index representing the probability that the respondent has a clinically relevant problem in sustained attention. Possible scores range from 0 to 100. Scores between 40 and 60 are considered inconclusive while scores above 60 indicate that the child exhibits inattentiveness.
Time Frame: Baseline, Month 6
Population: The analysis includes participants who completed the assessment at the specified study visit. Some participants attended a study visit but did not complete the CPT-II.
Measure: Mean (Standard Deviation); unit: Confidence Index
Arm/Group | Lamotrigine | Oxcarbazepine | Levetiracetam
Number analyzed (Participants) | 24 | 26 | 20
Confidence Index
  Baseline | 58.4 (20.0) | 56.7 (21.6) | 56.9 (23.9)
  After 6 months of treatment: number analyzed (Participants) | 17 | 22 | 14
  After 6 months of treatment | 58.1 (23.2) | 54.2 (21.7) | 54.0 (24.4)

2. Secondary Outcome: Child Behavior Checklist
Description: The Child Behavior Checklist is a measure of specific behavioral and emotional problems are rated by the child's parent or guardian. The Child Behavior Checklist examines three domains (Social Functioning, Mood and Anxiety Symptoms, and Externalizing Symptoms) by assessing 118 problem items that describe specific behavioral and emotional problems. Respondents indicate how accurately the statements describe the child by selecting from options on a 3-point Likert-type scale (0=Not True, 1= Somewhat or Sometimes True, or 2=Very True or Often True). Total raw scores are converted to t-scores with a mean of 50 and standard deviation of 10. A t-score of 67 or greater is considered to be in the clinical range for problematic behavior.
Time Frame: Baseline, Month 6
Population: The analysis includes participants who completed the assessment at the specified study visit. Some participants attended a study visit but did not complete the Child Behavior Checklist.
Measure: Mean (Standard Deviation); unit: t-scores
Arm/Group | Lamotrigine | Oxcarbazepine | Levetiracetam
Number analyzed (Participants) | 22 | 26 | 18
t-scores
  Baseline | 37.6 (9.9) | 39.8 (10.2) | 38.2 (10.3)
  After 6 months of treatment: number analyzed (Participants) | 16 | 21 | 12
  After 6 months of treatment | 37.5 (9.6) | 36.7 (11.1) | 33.3 (9.1)

3. Other Pre Specified Outcome: Wechsler Intelligence Scale for Children-IV Processing Speed
Description: Coding and Symbol Search subtests from the Wechsler Intelligence Scale for Children (WISC)-IV are measures of processing speed and combine to form the Processing Speed Index. Processing speed refers to how quickly the child understands and responds to information. Coding presents children with a row of boxes containing a numeral in the top line and a symbol in the bottom line with the task of copying the symbol corresponding to each numeral as quickly as possible in 120 seconds. In Symbol Search, children are given rows of symbols and target symbols and are asked to mark whether or not the target symbols appear in each row as quickly as possible during 120 seconds. Composite scores compare the test-taker to peers with a mean score of 100 and a standard deviation of 15. Possible scores range from 40 to 160 with higher scores indicating increased processing speeds. Scores between 85 and 115 are considered average, with 2/3 of test takers falling between these values.
Time Frame: Baseline, Month 3, Month 6
Population: The analysis includes participants who completed the assessment at the specified study visit. Some participants attended a study visit but did not complete the WISC-IV.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lamotrigine | Oxcarbazepine | Levetiracetam
Number analyzed (Participants) | 23 | 27 | 19
units on a scale
  Baseline | 87.8 (12.1) | 97.9 (15.5) | 102.1 (12.3)
  After 3 months of treatment: number analyzed (Participants) | 23 | 18 | 14
  After 3 months of treatment | 95.7 (16.7) | 90.4 (12.7) | 96.9 (14.0)
  After 6 months of treatment: number analyzed (Participants) | 15 | 23 | 12
  After 6 months of treatment | 97.3 (20.8) | 101.22 (19.1) | 102.6 (13.8)

4. Other Pre Specified Outcome: Story Memory
Description: Story Memory will be measured at baseline with the Children's Memory Scale (CMS) and then with the Wide Range Assessment of Memory and Learning-2 (WRAML-2) at the 6 month follow up visit. Two different tests are used to avoid practice effects in memory assessment associated with repeated assessments using the same stimulus material. The Story Memory sub-test of the CMS and the WRAML-2 Story Memory are measures of prose passage recall. Stories are read to the subject for recall, with different stories presented based upon participant age. Scores are converted to percentile ranks for both measurements of story memory. Possible scores can fall between the 1st and 99th percentile and higher values indicate better performance with story recall. Values between the 9th and 25 percentiles are considered "low average", values between the 25th and 75th percentiles are "average", while values between the 75th and 91st percentile are "high average".
Time Frame: Baseline, Month 6
Population: The analysis includes participants who completed the assessment at the specified study visit. Some participants attended a study visit but did not complete the Story Memory measurement.
Measure: Mean (Standard Deviation); unit: percentiles
Arm/Group | Lamotrigine | Oxcarbazepine | Levetiracetam
Number analyzed (Participants) | 22 | 26 | 20
percentiles
  Baseline (CMS) | 29.6 (16.2) | 31.2 (17.0) | 29.4 (12.2)
  After 6 months of treatment (WRAML-2): number analyzed (Participants) | 15 | 23 | 13
  After 6 months of treatment (WRAML-2) | 23.1 (13.9) | 26.1 (13.7) | 26.5 (9.3)

5. Other Pre Specified Outcome: Symbol Digit Modalities Test
Description: Symbol Digit Modalities Test (SDMT) is a test of graphomotor speed using numbers as the response rather than copying symbols, and is timed at 90 seconds. The SDMT is designed for people who are 8 years of age and older and detects brain dysfunction as well as measures function over time. Possible total scores range from 0 to 110; where 110 indicates that all values were entered within the 90 second limit. An increase between initial and retest scores indicates that the respondent is correctly matching numbers to symbols at a faster speed. The SDMT was administered at the Month 3 and Month 6 visits for this study.
Time Frame: Month 3, Month 6
Population: The analysis includes participants who completed the assessment at the specified study visit. Participants who were 8 years old or older were eligible to complete the Symbol Digit Modalities Test.
Measure: Mean (Standard Deviation); unit: number of correct responses
Arm/Group | Lamotrigine | Oxcarbazepine | Levetiracetam
Number analyzed (Participants) | 10 | 15 | 9
number of correct responses
  After 3 months of treatment: number analyzed (Participants) | 10 | 13 | 9
  After 3 months of treatment | 25.9 (10.3) | 28.5 (10.3) | 23.0 (9.4)
  After 6 months of treatment: number analyzed (Participants) | 9 | 15 | 6
  After 6 months of treatment | 26.4 (11.3) | 30.4 (12.3) | 28.3 (8.6)

6. Other Pre Specified Outcome: Grooved Pegboard
Description: The Grooved Pegboard assesses fine motor speed and dexterity. The participant fits keyhole-shaped pegs into similarly shaped holes on a square board. The pegs, which have an edge along one side, must be rotated to match the holes before they can be inserted. The scores represent the number of seconds it took for the participant to correctly insert the pegs into the require number of grooves, using their dominant hand.
Time Frame: Baseline, Month 6
Population: The analysis includes participants who completed the assessment at the specified study visit. Some participants attended a study visit but did not complete the Grooved Pegboard task.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Lamotrigine | Oxcarbazepine | Levetiracetam
Number analyzed (Participants) | 21 | 26 | 20
Seconds
  Baseline | 99.9 (24.8) | 96.3 (24.0) | 114.2 (36.2)
  After 6 months of treatment: number analyzed (Participants) | 15 | 23 | 13
  After 6 months of treatment | 90.3 (34.7) | 90.1 (24.2) | 94.9 (19.7)

7. Other Pre Specified Outcome: The Number of Participants With a Positive Response on the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: Suicidal behaviors and suicidal ideation were assessed through an interview using the Columbia-Suicide Severity Rating Scale (C-SSRS). The C-SSRS guides interviewers to ask a series of simple questions in order to identify people at risk for suicide, as well as the severity and urgency of suicidal thoughts and behaviors. The Children's Baseline/Screening C-SSRS was used at the initial study visit while the Children's Since Last Visit C-SSRS was used for subsequent study visits. Any responses of "yes" to the C-SSRS questions are considered a positive response, indicating that the participant is experiencing thoughts of suicide or has exhibited suicidal behaviors.
Time Frame: Baseline, Month 3, Month 6
Population: The analysis includes participants who completed the assessment at the specified study visit. Some participants attended a study visit but did not complete the C-SSRS.
Measure: Count of Participants; unit: Participants
Arm/Group | Lamotrigine | Oxcarbazepine | Levetiracetam
Number analyzed (Participants) | 23 | 27 | 20
Participants
  Baseline | 0 | 0 | 0
  After 3 months of treatment: number analyzed (Participants) | 20 | 21 | 15
  After 3 months of treatment | 0 | 0 | 0
  After 6 months of treatment: number analyzed (Participants) | 20 | 21 | 15
  After 6 months of treatment | 0 | 0 | 0

8. Other Pre Specified Outcome: Youth Self Report
Time Frame: 6 months
Population: As this study was terminated early, the scoring algorithm was not programmed for this outcome measure.
Arm/Group | Lamotrigine | Oxcarbazepine | Levetiracetam
Number analyzed (Participants) | 0 | 0 | 0

9. Other Pre Specified Outcome: Affective Reactivity Scale
Description: The Affective Reactivity Scale is a 7-item survey completed by the child participants which asks questions concerning their level of agreement with statements about anger and irritability. Respondents select between "not true" (scored as 0), "somewhat true" (scored as 1), and "certainly true (scored as 2). Total scores range from 0 to 14 with higher values indicating increased feelings of annoyance and anger.
Time Frame: Baseline, Month 3, Month 6
Population: The analysis includes participants who completed the assessment at the specified study visit. Some participants attended a study visit but did not complete the Affective Reactivity Scale.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lamotrigine | Oxcarbazepine | Levetiracetam
Number analyzed (Participants) | 24 | 27 | 21
units on a scale
  Baseline | 9.2 (2.5) | 8.6 (2.7) | 8.6 (2.2)
  After 3 months of treatment: number analyzed (Participants) | 21 | 23 | 15
  After 3 months of treatment | 8.8 (2.5) | 8.5 (2.0) | 10.3 (3.1)
  After 6 months of treatment: number analyzed (Participants) | 16 | 24 | 15
  After 6 months of treatment | 8.8 (3.0) | 8.2 (2.7) | 10.3 (3.2)

10. Other Pre Specified Outcome: Pediatric Neuro-QOL Score
Description: The Pediatric Neuro-QOL is a Quality of Life instrument developed in conjunction with NIH with a pediatric specific form utilized in this protocol. Pediatric Neuro-QOL assesses the domains of Anger, Anxiety, Cognition, Depression, Fatigue, Pain, Social Relations, and Stigma. Each domain has 8 to 10 items and respondents indicate how often they experienced feelings and circumstances related to each domain on a scale of 1 to 5 (such as 1=never, 2=almost never, 3=sometimes, 4=often, 5=almost always). Higher values indicate increased difficulty for most of the scales but this pattern is reversed for two of the domains. Raw scores are rescaled to standardized scores with a mean of 50 and a standard deviation of 10. Higher values for the standardized scores indicate more problematic characteristics while scores below 50 indicate that the child is experiencing less trouble in the domains measured by the Pediatric Neuro-QOL.
Time Frame: Baseline, Month 6
Population: The analysis includes participants who completed the assessment at the specified study visit. This survey was completed by children aged 10 and older.
Measure: Mean (Standard Deviation); unit: t-scores
Arm/Group | Lamotrigine | Oxcarbazepine | Levetiracetam
Number analyzed (Participants) | 14 | 15 | 11
t-scores
  Baseline | 37.0 (6.0) | 39.9 (9.6) | 38.8 (5.6)
  After 6 months of treatment: number analyzed (Participants) | 8 | 14 | 7
  After 6 months of treatment | 36.7 (8.2) | 35.2 (5.2) | 36.9 (5.3)

11. Other Pre Specified Outcome: Parenting Stress Inventory Short Form (PSI-4-SF)
Description: The Parenting Stress Inventory-4-Short Form is a 36 item questionnaire, completed by the parent/guardian, designed to evaluate parenting and family characteristics based upon child characteristics (behavioral and emotional problems), parent characteristics, and situational/demographic life stress. Respondents indicate the degree to which they agree with a variety of statements by selecting 1=strongly agree, 2=agree, 3=not sure, 4=disagree, or 5=strongly disagree. Raw scores range from 36 to 180 and higher scores are associated with higher parental stress.
Time Frame: Baseline, Month 6
Population: The analysis includes participants who completed the assessment at the specified study visit. Some parents attended a study visit but did not complete the PSI-4-SF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lamotrigine | Oxcarbazepine | Levetiracetam
Number analyzed (Participants) | 22 | 22 | 20
units on a scale
  Baseline | 138.2 (21.0) | 138.3 (17.5) | 143.9 (20.4)
  After 6 months of treatment: number analyzed (Participants) | 17 | 22 | 12
  After 6 months of treatment | 147.4 (20.9) | 137.6 (24.3) | 146.8 (22.3)

12. Other Pre Specified Outcome: Pediatric Inventory for Parents
Description: The Pediatric Inventory for Parents consists of 42 items involving communication, medical care, emotional disturbance, and change in role function. Parents respond to a list of difficult events (such as "difficulty sleeping") that are often experienced by parents of children who are seriously ill. Parents indicated how frequently an event occurred by selecting 1=Never, 2=Rarely, 3=Sometimes, 4=Often, or 5=Very often. Raw score values range from 4 to 210 with higher scores indicating increased frequency of difficult events.
Time Frame: Baseline, Month 6
Population: The analysis includes participants who completed the assessment at the specified study visit. Some parents attended a study visit but did not complete the Pediatric Inventory for Parents.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lamotrigine | Oxcarbazepine | Levetiracetam
Number analyzed (Participants) | 24 | 25 | 21
units on a scale
  Baseline | 93.0 (21.5) | 98.4 (33.2) | 91.1 (29.9)
  After 6 months of treatment: number analyzed (Participants) | 17 | 21 | 13
  After 6 months of treatment | 74.2 (20.3) | 76.5 (32.0) | 74.8 (17.6)

ADVERSE EVENTS:
Time Frame: Information about adverse events experienced by participants was collected from the time the participant began taking the randomized study drug through 30 days after the last study visit.
Description: An adverse event (AE) is an unfavorable and unintended diagnosis, sign, symptom, or disease temporarily associated with the study intervention. Serious adverse events (SAEs) are untoward medical occurrence resulting in death, are life-threatening, require or prolong hospitalization, cause disability/incapacity, result in birth defects, or represent other significant hazards. For this study, elective hospitalizations unrelated to epilepsy will not be considered SAEs.
Arm/Group | Lamotrigine | Oxcarbazepine | Levetiracetam
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/27 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/27 | 0/21
Other Adverse Events (participants affected / at risk) | 0/24 | 0/27 | 0/21

LIMITATIONS AND CAVEATS:
The study was terminated early due to inability to meet enrollment goals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes